CLINICAL TRIAL: NCT02857478
Title: To Assess the Safety of a Sunscreen Product,BAY 987519, Bayer Sponsored, CC Products
Brief Title: Supervised Outdoor-Use Test to Assess the Safety of a Sunscreen C-Spray on Sport Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 18317
Record Dates: First submitted 2016-08-03; First posted 2016-08-05 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Sunscreen Agents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Safety of a Sunscreen product (Experimental): Sunscreen product safety evaluation under supervised out-door conditions on sport users.
  Interventions: Drug: BAY 987519, SPF 50, Y51-002; Drug: BAY 987519, SPF 50, P04-147

INTERVENTIONS:
Drug: BAY 987519, SPF 50, Y51-002 — Sufficient amount to cover all exposed skin liberally two times - approximately 240 min.
Drug: BAY 987519, SPF 50, P04-147 — Sufficient amount to cover all exposed skin liberally two times - approximately 240 min.

SUMMARY:
The objective of this study was to assess the safety and appropriateness of a sunscreen product for use on sport users, under supervised outdoor-use conditions. The study was conducted under the supervision of a Board-Certified Dermatologist at an outdoor, chlorinated swimming pool facility.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged 18 to 65 years
* No actinic keratosis, skin cancer, psoriasis, eczema, or any other acute or chronic skin conditions
* Must not have visible erythema, blistering or peeling that would indicate recent sunburn
* Must not have asthma. Must not be undergoing therapy with system or topical corticosteroids, anti-inflammatories or antihistamine agents
* Must not be taking any medication in which exposure to the sun is contraindicated
* Must be willing to obey all rules of the test facility

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2015-06-27 (Actual); Primary Completion 2015-06-28 (Actual); Study Completion 2015-06-28 (Actual)

PRIMARY OUTCOMES:
Evaluation of Erythema as graded on a 5 point scale. | approximately 24 hours
Evaluation of AEs, including eye stinging | approximately 24 hours
  Reported as product related or likely product related by the investigator or trained designee

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- St. Petersburg, Florida, United States